CLINICAL TRIAL: NCT04345068
Title: A Pilot Study of Calm for Cancer Patient Sleep Disturbance
Brief Title: Calm for Cancer Sleep Disturbance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Arizona State University (Other)
Collaborators: The University of Texas Health Science Center at San Antonio (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: STUDY00011444
Record Dates: First submitted 2020-04-09; First posted 2020-04-14 (Actual); Last update posted 2022-02-25 (Actual); Status verified 2022-02

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Who Masked: Participant
Masking Description: The participants will be blinded as to which group is receiving the intervention being assessed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Calm Meditation (Experimental): The intervention will be 8-weeks in duration and will consist of a series of pre-approved meditation classes. Patients will be asked to participate in at least 10 min/day of meditation (i.e., ~70 min/week). Week 1-4 will consist of the "7 Days of Calm" followed by the "21 Days of Calm", which are introductory courses offered by Calm and provide basic, introductory meditation classes for beginners. Weeks 5-8 will consist of patients participating in the "Daily Calm" that Calm provides, consisting of 10-12 min meditation classes that have a unique focus each day. Patients will be instructed to participate in at least 10 min/day of meditation, but will be encouraged to do more if they can.
  Interventions: Behavioral: Calm Meditation Mobile App
- Health Education Podcast (Active Comparator): The control group will serve as an active control group and will be matched for time and attention to the intervention group. Participants assigned to the control group will be asked to listen to/view 10-min/day (i.e., ~70 min/week) of health education podcasts via a smartphone app. Topics covered in the health education control vary and will be aimed at providing useful and informative health-related information pertinent to cancer patients. The podcast app was developed by an independent app developer, and it was designed to mirror the type of functionality that the Calm app offers its users.
  Interventions: Behavioral: Health Education Podcast Mobile App

INTERVENTIONS:
Behavioral: Calm Meditation Mobile App — The Calm app is downloadable by participants onto their smartphone. The Calm app is used to deliver the meditation intervention to experimental group participants.
  Arms: Calm Meditation
Behavioral: Health Education Podcast Mobile App — The health education podcast mobile app mirrors the intervention group's app experience, but provides educational content via podcasts as an active comparator.
  Arms: Health Education Podcast

SUMMARY:
Cancer and cancer treatment often lead patients and survivors to experience a host of chronic symptoms, of which sleep disturbances are a major concern. Smartphone-based meditation via an already-developed app (i.e., Calm) is a unique and novel way of providing a potentially helpful symptom-management strategy to cancer patients and survivors. Our hypothesis is that cancer patients/survivors using the Calm smartphone app for eight weeks will see improved sleep disturbance (primary outcome) as well as anxiety, depression, pain intensity, global health, quality of life, emotional regulation, and mindfulness when compared to a time and attention-matched health education podcast control group. Cancer patients/survivors (n=300) will be randomly assigned to an intervention or control group for eight weeks, with study outcome measurement occurring at baseline, post-intervention (i.e., week eight), and follow-up (i.e., week 20).

DETAILED DESCRIPTION:
Cancer patients and survivors struggle with chronic symptom burden, including sleep disturbance, fatigue, depressive symptoms, and anxiety, among others. Sleep disturbance is one of the most common complaints among cancer patients and survivors (reported in as many as 85% of cancer patients and survivors, depending on the type of cancer), but is often not fully addressed by pharmacologic intervention alone. Therefore, cancer patients and survivors often turn to non-pharmacologic approaches.

Currently, cognitive behavioral therapy for insomnia (CBT-I) is the most available, evidence-based, non-pharmacologic treatment strategy to manage sleep disturbances in cancer patients and survivors. However, this treatment modality is time-consuming and intensive, requiring patients to frequently meet in-person with therapists and physicians at sites/clinics. This approach may not be sustainable in the long term, as cancer patients often report barriers to attending in-person interventions, including fatigue, transportation, and scheduling difficulties. Although remote delivery of CBT-I has been suggested as an alternative,1 only a single pilot study has investigated this possibility. The pilot study delivered CBT-I via a mobile app, but was limited by the small sample size (n=19) and no control group. Further research is needed testing the delivery of efficacious, non-pharmacologic interventions remotely to cancer patients and survivors for the management of sleep disturbance.

Smartphones, due to their increasing ubiquity among cancer patients and survivors, offer a novel medium through which to deliver non-pharmacologic sleep-management interventions. In a recent survey of 1,300 cancer patients, 71% reported owning a mobile smartphone. A 2018 survey of 631 cancer patients demonstrated that 74% regularly use a smartphone, and 39% expressed an interest in supportive care information via mobile apps. Meditation is a non-pharmacologic intervention that has a growing body of literature to document its benefits for sleep in cancer patients, and it is a less time-consuming and resource-intensive strategy when compared to CBT-I. Further research needs to examine the potential efficacy of meditation as an efficacious non-pharmacologic strategy for the self-management of sleep disturbances.

The investigators have successfully delivered meditation to hematological cancer patients previously via the Calm app with moderate effects demonstrated on sleep disturbance. However, more research is needed to test the preliminary effects of smartphone-based meditation among cancer patients for sleep disturbance as compared to an active control group. In the proposed study, the investigators will recruit a national sample of cancer patients and survivors (N=300) within two years of cancer diagnosis, to pilot test an eight-week smartphone-based meditation intervention (i.e., Calm; n=150) on sleep disturbance (primary outcome) as compared to a smartphone-based health education podcast control group (n=150). The investigators will aim to recruit 50% men into the study.

STUDY OBJECTIVES

Objective 1: Explore the preliminary effects of eight weeks of daily meditation delivered using the Calm app on sleep disturbance in cancer patients and survivors within two years of diagnosis as compared to a smartphone-based podcast control group.

The primary hypothesis for this objective is that those in the Calm group will experience improvements in sleep disturbance greater than those experienced by the podcast control group at eight weeks.

Objective 2: Explore the preliminary effects of eight weeks of daily meditation delivered using the Calm app on cancer patients and survivors within two years of diagnosis on anxiety, depression, pain intensity, global health, quality of life, emotional regulation, and mindfulness as compared to a smartphone-based podcast control group.

The primary hypothesis for this objective is that those in the Calm app group will experience improvements in anxiety, depression, pain intensity, global health, quality of life, emotional regulation, and mindfulness greater than those experienced by the podcast control group at eight weeks.

Exploratory Objective 3: Explore the sustained effects of meditation delivered using the Calm app on cancer patients and survivors (i.e., 12-week follow-up).

The primary hypothesis for this objective is that those in the Calm app group will experience improvements across outcomes compared to baseline that are sustained at 20 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Have a cancer diagnosis within the past 2 years
* self-identify as sleep disturbed (Pittsburgh Sleep Quality Index score of >5 indicating moderate sleep disturbance)
* own a mobile smartphone (iPhone with iOS 9.0 or later or an Android 4.1 or later)
* willing to download a mobile app
* able to read and understand English
* aged 18 years or older
* willing to be randomized to one of two groups
* no change in pharmacologic therapy over the past two weeks
* no change in sleep medication use (if any) over the past six weeks

Exclusion Criteria:

* meditation or meditative movement practice (i.e., yoga, tai chi, qigong) of greater than or equal to 60 min/month in the past six months
* use of any consumer-based meditation app
* reside outside of the United States
* any planned change in pharmacologic therapy or planned stem cell transplant during the study interval (i.e., 20 weeks)
* self-reported sleep-disordered breathing and/or sleep movement disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2020-08-01 (Actual); Primary Completion 2021-06-01 (Actual); Study Completion 2021-06-01 (Actual)

PRIMARY OUTCOMES:
Change in Sleep Disturbance | Change from baseline to mid-point (week 4), to post-intervention (week 8)
  Sleep Disturbance will be measured with the NIH PROMIS Sleep Disturbance Adult Short Form. A higher score indicates more of the concept being measured.

SECONDARY OUTCOMES:
Change in Anxiety | Change from baseline to mid-point (week 4), to post-intervention (week 8)
  Anxiety will be measured with the NIH PROMIS Anxiety Short Form. A higher score indicates more of the concept being measured.
Change in Depression | Change from baseline to mid-point (week 4), to post-intervention (week 8)
  Depression will be measured with the NIH PROMIS Depression Adult Short Form. A higher score indicates more of the concept being measured.
Change in Pain Intensity | Change from baseline to mid-point (week 4), to post-intervention (week 8)
  Pain Intensity will be measured with the NIH PROMIS Pain Intensity Adult Short Form. A higher score indicates more of the concept being measured.
Change in Global Health | Change from baseline to mid-point (week 4), to post-intervention (week 8)
  Global Health will be measured with the NIH PROMIS Global Health. A higher score indicates more of the concept being measured.
Overall Quality of Life | Change from baseline to mid-point (week 4), to post-intervention (week 8)
  Overall Quality of Life will be measured with the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC-QLQC30). A higher score indicates more of the concept being measured.
Emotional Regulation | Change from baseline to mid-point (week 4), to post-intervention (week 8)
  Emotional Regulation will be measured with the Difficulties in Emotion Regulation Scale Short Form. This form is an 18-item measure used to identify emotional regulation issues in adults. The measure covers 4 dimensions of emotional regulation: awareness and understanding of emotions; acceptance of emotions; the ability to engage in goal-directed behavior and refrain from impulsive behavior when experiencing negative emotions; and access to emotion regulation strategies perceived as effective. The measure has six subscales: Nonacceptance of emotional responses, difficulty engaging in goal-directed behavior, impulse control difficulties, lack of emotional awareness, limited access to emotion regulation strategies, and lack of emotional clarity. A higher score indicates greater difficulties in emotional regulation.
Mindfulness | Change from baseline to mid-point (week 4), to post-intervention (week 8)
  Mindfulness will be measured with the Mindful Attention Awareness Scale (MAAS). The MAAS is a 15-item scale designed to assess a core characteristic of dispositional mindfulness. Higher scores reflect higher levels of dispositional mindfulness.

OTHER OUTCOMES:
Sustained Effects on Sleep Disturbance | Change from post-intervention (week 8) to follow-up (week 20)
  Sleep Disturbance will be measured with the NIH PROMIS Sleep Disturbance Adult Short Form. A higher score indicates more of the concept being measured.
Sustained Effects on Depression | Change from post-intervention (week 8) to follow-up (week 20)
  Depression will be measured with the NIH PROMIS Depression Adult Short Form. A higher score indicates more of the concept being measured.
Sustained Effects on Anxiety | Change from post-intervention (week 8) to follow-up (week 20)
  Anxiety will be measured with the NIH PROMIS Anxiety Short Form. A higher score indicates more of the concept being measured.
Sustained Effects on Pain Intensity | Change from post-intervention (week 8) to follow-up (week 20)
  Pain Intensity will be measured with the NIH PROMIS Pain Intensity Adult Short Form. A higher score indicates more of the concept being measured.
Sustained Effects on Global Health | Change from post-intervention (week 8) to follow-up (week 20)
  Global Health will be measured with the NIH PROMIS Global Health. A higher score indicates more of the concept being measured.
Sustained Effects on Overall Quality of Life | Change from post-intervention (week 8) to follow-up (week 20)
  Overall Quality of life will be measured with the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC-QLQC30). A higher score indicates more of the concept being measured.
Sustained Effects on Emotional Regulation | Change from post-intervention (week 8) to follow-up (week 20)
  Emotional Regulation will be measured with the Difficulties in Emotion Regulation Scale Short Form. This form is an 18-item measure used to identify emotional regulation issues in adults. The measure covers 4 dimensions of emotional regulation: awareness and understanding of emotions; acceptance of emotions; the ability to engage in goal-directed behavior and refrain from impulsive behavior when experiencing negative emotions; and access to emotion regulation strategies perceived as effective. The measure has six subscales: Nonacceptance of emotional responses, difficulty engaging in goal-directed behavior, impulse control difficulties, lack of emotional awareness, limited access to emotion regulation strategies, and lack of emotional clarity. A higher score indicates greater difficulties in emotional regulation.
Sustained Effects on Mindfulness | Change from post-intervention (week 8) to follow-up (week 20)
  Mindfulness will be measured with the Mindful Attention Awareness Scale (MAAS). The MAAS is a 15-item scale designed to assess a core characteristic of dispositional mindfulness. Higher scores reflect higher levels of dispositional mindfulness.

CONTACTS AND LOCATIONS:
Locations (1):
- Arizona State University, Phoenix, Arizona, United States

IPD SHARING:
Plan to Share IPD: No